CLINICAL TRIAL: NCT02191228
Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Single and Multiple 5 mg Doses of Linagliptin Tablets in Patients With Different Degrees of Renal Impairment in Comparison to Subjects With Normal Renal Function in a Monocentric, Open, Parallel-group, Phase I Trial
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Single and Multiple Doses of Linagliptin Tablets in Patients With Different Degrees of Renal Impairment in Comparison to Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1218.26
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-06

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency | interventions — Linagliptin

ARMS (7):
- Group 1 (Experimental): Linagliptin in subjects with normal renal function
  Interventions: Drug: Linagliptin - Multiple dose
- Group 2 (Experimental): Linagliptin in patients with mild renal insufficiency (RI)
  Interventions: Drug: Linagliptin - Multiple dose
- Group 3 (Experimental): Linagliptin in patients with moderate RI
  Interventions: Drug: Linagliptin - Multiple dose
- Group 4 (Experimental): Linagliptin in patients with severe RI
  Interventions: Drug: Linagliptin - single dose
- Group 5 (Experimental): Linagliptin in patients with end-stage renal disease (ESRD)
  Interventions: Drug: Linagliptin - single dose
- Group 6 (Experimental): Linagliptin in patients with severe RI and Type 2 diabetes mellitus (T2DM)
  Interventions: Drug: Linagliptin - Multiple dose
- Group 7 (Experimental): Linagliptin in patients with normal renal function and T2DM
  Interventions: Drug: Linagliptin - Multiple dose

INTERVENTIONS:
Drug: Linagliptin - single dose
  Arms: Group 4; Group 5
Drug: Linagliptin - Multiple dose
  Arms: Group 1; Group 2; Group 3; Group 6; Group 7

SUMMARY:
The main objective of this study was to assess the effect of normal and impaired renal function on the safety, pharmacokinetics, and pharmacodynamics of linagliptin following oral administration of 5 mg daily for 7 days (Groups 1 to 3), 5 mg daily for 10 days (Groups 6 and 7), or as a single dose (Groups 4 and 5)

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with normal renal function, defined as a Creatinine Clearance (CrCl) of >80 mL/min on screening (Group 1) , or male or female patients with Type 2 diabetes mellitus (T2DM) and normal renal function, defined as a CrCl of >80 mL/min on screening (Group 7)
* Male or female patients with Renal impairment (RI), determined by the value of CrCl on Screening estimated according to the Cockcroft-Gault formula. Patients were classified into groups by their CrCl values:

  * Mild RI: CrCl>50 to ≤80 mL/min (Group 2)
  * Moderate RI: CrCl>30 to ≤50 mL/min (Group 3)
  * Severe RI: CrCl≤30 mL/min (Group 4)
  * End-stage renal disease (ESRD): CrCl≤30 mL/min, requiring hemodialysis (Group 5)
  * T2DM and severe RI: CrCl≤30 mL/min (Group 6)
* Age 18 to 80 years
* BMI 18 to 40 kg/m2, and minimum body mass of at least 45 kg for females
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP) and the local legislation

Exclusion Criteria:

Participants (with or without RI) who met any of the following criteria were not included in this trial:

* Relevant gastrointestinal tract surgery (except appendectomy, cholecystectomy, or herniotomy)
* Diseases of the central nervous system, such as epilepsy, seizures, relevant neurological disorders, or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts; systolic blood pressure <100 or >160 mm Hg, diastolic blood pressure <60 or >100 mm Hg, pulse rate <50 or >100 1/min
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergies) that were deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (>24 h) within at least one month prior to study start, or planned intake of study medication within ≤10 half-lives of administration of another medication. Medications that patients with RI were currently taking for treatment of renal disease were not included under this criterium.
* Use of medications during the trial or within 10 days prior to administration of study medication that might reasonably influence the results of the trial, based on knowledge at the time of protocol preparation. Co-medications known to inhibit or induce P-glycoprotein or CYP3A were not allowed. Inhibitors of P-glycoprotein or CYP3A include protease inhibitors (such as ritonavir, lopinavir, nelfinavir); azole antimycotics, (itraconazole, ketoconazole, miconazole); macrolide antibiotics, (clarithromycin, erythromycin); amiodarone, cimetidine, diltiazem, fluvoxamine, mibefradil, nefazodone, verapamil, tacrolimus, quinidine, reserpine, and cyclosporine A. Inducers of P-gp or CYP3A include carbamazepine, phenobarbital, phenytoin, rifabutin, rifampin, St. John's Wort and troglitazone. In uncertain cases, a case-by-case decision was made after consultation with the sponsor.
* Participation in a previous trial with an investigational drug within 2 months of study start if the previous trial was a multiple dose study, or within 1 month of study start if the previous trial was a single dose study
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking when confined to the study site on trial days
* Alcohol abuse (more than 60 g/day in males or more than 40 g/day in females)
* Drug abuse, in the investigator's judgment, based on review of the participant's history and urine screening for abused substances
* Veins unsuited for intravenous puncture on either arm (e.g. veins which were difficult to locate, access or puncture, veins with a tendency to rupture during or after puncture)
* Blood donation (more than 100 mL within 4 weeks prior to administration of study medication or during the trial)
* Excessive physical activities (within 48 h prior to start of the trial or during the trial)
* Any laboratory value outside the reference range that was of clinical relevance (exceptions were in patients with RI who had abnormal renal function tests or deviations of clinical laboratory values that were related to renal impairment)
* Inability to comply with the dietary regimen of study centre
* Inability to understand and comply with protocol requirements, instructions and protocol-stated restrictions

For female patients

* Pregnancy
* Positive pregnancy test (human chorionic gonadotropin (β HCG) in urine))
* No adequate contraception in women of childbearing potential (adequate contraception was considered to be sterilisation, use of an intrauterine device, or use of oral contraception along with a barrier method)
* Lactation period

Subjects with normal renal function (Group 1) and subjects with T2DM and normal renal function (Group 7) who met the following criterium were not included in this trial:

* Significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders as judged by the investigator

Patients with RI who met any of the following criteria were not included in this trial:

* Moderate and severe concurrent liver function impairment (for example, due to hepatorenal syndrome)
* Patients with significant diseases other than renal impairment were excluded. A significant disease was defined as a disease which in the opinion of the investigator put the patient at risk during participation in the study, could influence the results of the study, could influence the patient's ability to participate in the study, or was an unstable condition. Patients with diabetes (for Groups 1 to 5) or hypertension could be included in the trial if the disease was not significant according to these criteria.
* Haemoglobin <8 g/dL, indicating severe anaemia of renal origin (use of erythropoietin was allowed to maintain haematocrit)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-04; Primary Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
AUCτ,ss (area under the concentration time curve of the analyte in plasma over the time interval from 0 to 24h after the last dose at steady state) - multiple dose groups | up to 480 hours
Cmax,ss (maximum concentration of the analyte in plasma at steady state) - multiple dose groups | up to 480 hours
AUC0-24 (area under the concentration time curve of the analyte in plasma over the time interval from 0 to 24h after the first dose) - single dose groups | up to 24 hours
Cmax (maximum concentration of the analyte in plasma) - single dose groups | up to 264 hours

SECONDARY OUTCOMES:
tmax,(ss) (time from last dosing to maximum concentration of the analyte in plasma after the first dose or at steady state) - multiple dose groups | up to 480 hours
C24,(ss) (concentration of the analyte in plasma at steady state after administration of the first or last dose at the end of the dosing interval) - multiple dose groups | up to 480 hours
λz,(ss) (terminal rate constant in plasma after single dose/at steady state) - multiple dose groups | up to 480 hours
t1/2,(ss) (terminal half-life of the analyte in plasma after single dose/at steady state) - multiple dose groups | up to 480 hours
MRTpo,(ss) (mean residence time of the analyte in the body after single dose/at steady state after oral administration) - multiple dose groups | up to 480 hours
CL/F,(ss) (apparent clearance of the analyte in the plasma after extravascular administration after single dose/at steady state) - multiple dose groups | up to 480 hours
Vz/F,(ss) (apparent volume of distribution during the terminal phase λz after single dose/at steady state following extravascular administration) - multiple dose groups | up to 480 hours
AUC0-∞ (area under the concentration time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity after single dose in severely impaired or end stage renal disease (ESRD) patients) | up to 264 hours
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point after single dose in severely impaired or ESRD patients) | up to 264 hours
%AUCtz-∞ (percentage of area under the concentration-time curve of the analyte in plasma over the time interval from the time of the last quantifiable data point extrapolated to infinity after single dose in severely impaired or ESRD patients) | up to 264 hours
Assessment of Plasma protein binding | predose Day 1
Model-derived AUCτ,ss in severely impaired or ESRD patients | up to 264 hours
Model-derived Cmax,ss in severely impaired or ESRD patients | up to 264 hours
Change in Dipeptidyl peptidase IV (DPP-4) activity in plasma | up to 480 hours
Number of patients with abnormal findings in physical examination | up to day 32
Number of patients with clinically significant changes in vital signs | up to day 32
Number of patients with abnormal changes 12-lead ECG (electrocardiogram) | up to day 32
Number of patients with abnormal changes in laboratory parameters | up to day 32
Number of patients with adverse events | up to 53 days
Assessment of tolerability by investigator on a 4-point scale | up to 480 hours
AUC0-24 (area under the concentration time curve of the analyte in plasma over the time interval from 0 to 24h after the first dose) - multiple dose groups | up to 24 hours
Cmax (maximum concentration of the analyte in plasma) - multiple dose groups | up to 480 hours